CLINICAL TRIAL: NCT01114152
Title: A Phase I, Single Center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Intravenous AZD9742 in Healthy Male and Female Japanese Subjects
Brief Title: AZD9742 Single and Multiple Ascending Dose Study in Healthy Male and Female Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2690C00003
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: AZD9742; Japanese Healthy Volunteers; Phase I; Single and Multiple Ascending Dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dose level A, B, C and optional Dose level D and E: single administration and one to three times daily for 6 days (Japanese n=8)
  Interventions: Drug: AZD9742
- 2 (Placebo Comparator): placebo given (2 subjects in each dose group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9742 — IV Formulation
  Arms: 1
Drug: Placebo — IV Formulation
  Arms: 2

SUMMARY:
This is a Phase I randomized double-blind, placebo-controlled, single and multiple ascending dose study to assess the safety, tolerability and pharmacokinetics of AZD9742 in healthy male and female Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* female (non-childbearing potential)
* Body mass index (BMI) : 17 to 27 kg/m 2

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic, or renal disease or any otherHistory or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, physical examinations, clinical laboratory assessments, 12-lead ECG, digital ECG, telemetry) | collected prior to treatment, during treatment and follow-up for a total of 18-22 days

SECONDARY OUTCOMES:
Characterize the Pharmacokinetics of AZD9742 in blood and urine | PK-sampling during 14 pre-defined study days for PK profiling

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, M..D., Principal Investigator — California Clinical Trials; David Melnick, Study Director — AstraZeneca
Locations (1):
- Research Site, Glendale, California, United States